CLINICAL TRIAL: NCT02730455
Title: Multicenter, Double-Blind, Placebo-Controlled, Randomized, Parallel-Group, Dose-Ranging Study to Evaluate the Safety and Efficacy of Intravenous Natalizumab (BG00002) in Acute Ischemic Stroke
Brief Title: Safety and Efficacy of Intravenous Natalizumab in Acute Ischemic Stroke
Acronym: ACTION2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101SK202; 2015-004783-11 (EudraCT Number)
Record Dates: First submitted 2016-03-10; First posted 2016-04-06 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Natalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- natalizumab high dose (Experimental): Single IV (intravenous) dose natalizumab at baseline at one of two treatment windows, either within 9 hours of last known normal (LKN) or between 9-24 hours after LKN.
  Interventions: Drug: natalizumab
- natalizumab low dose (Experimental): Single IV (intravenous) dose natalizumab at baseline at one of two treatment windows, either within 9 hours of last known normal (LKN) or between 9-24 hours after LKN.
  Interventions: Drug: natalizumab
- Placebo (Experimental): Single dose of Placebo IV at baseline at one of two treatment windows, either within 9 hours of last known normal (LKN) or between 9-24 hours after LKN.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: natalizumab — Administered as specified in the treatment arm
  Other Names: BG00002
  Arms: natalizumab high dose; natalizumab low dose
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the clinical effects of natalizumab versus placebo in acute ischemic stroke on clinical measures of functional independence and activities of daily living. The secondary objective of the study is to explore dose and exposure response and the clinical treatment effects of natalizumab versus placebo in acute ischemic stroke on the following: measures of independence, activities of daily living, neurologic function, quality of life, cognition, and safety and tolerability

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of supratentorial acute ischemic stroke defined by LKN ≤24 hours prior to study treatment initiation.
* Score of 5 to 23 points, inclusive, on the NIHSS at Screening for subjects initiating treatment ≤9 hours from LKN. Note: NIHSS eligibility must be confirmed within 60 minutes prior to randomization.
* Score of 5 to 15 points, inclusive, on the NIHSS at Screening for subjects initiating treatment >9 to ≤24 hours from LKN. Note: NIHSS eligibility must be confirmed within 60 minutes prior to randomization.
* Prior to index stroke, patient was able to perform basic activities of daily living without assistance: dressing, eating, walking, bathing, and using the toilet.
* For those subjects who underwent a cranial MRI, there is at least 1 acute infarct with a diameter of ≥2 cm on baseline brain diffusion-weighted imaging.

Key Exclusion Criteria:

* Lacunar or isolated brainstem or cerebellar stroke based on clinical assessment and available acute imaging studies performed under the standard of care.
* Presence of acute intracranial hemorrhage on acute brain CT or MRI. However, petechial hemorrhages of ≤1 cm are not exclusionary.
* Severe stroke defined by imaging criteria based on either one of the following:
* Alberta Stroke Program Early CT (ASPECT) score of 0 to 4 based on head CT or
* Acute infarct volume on MRI diffusion weighed imaging greater than or equal to 70 mL
* Seizure at the onset of stroke.
* Known history of prior treatment with natalizumab.
* Known history of active viral hepatitis B or C.
* Signs and symptoms of active or acute infection.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (46):
- United States (16):
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainesville, Florida
  - Research Site, Fort Wayne, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Knoxville, Tennessee
- Germany (18):
  - Research Site, Altenburg
  - Research Site, Bad Neustadt/Saale
  - Research Site, Bamberg
  - Research Site, Bergisch Gladbach
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, Ludwigshafen
  - Research Site, Mannheim
  - Research Site, Minden
  - Research Site, Münster
  - Research Site, Trier
  - Research Site, Tübingen
  - Research Site, Ulm
- Spain (9):
  - Research Site, Albacete
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Valladolid
- United Kingdom (3):
  - Research Site, London, Greater London
  - Research Site, Harrow, Middlesex
  - Research Site, Stoke-on-Trent, Staffordshire

REFERENCES:
- [Derived] Elkind MSV, Veltkamp R, Montaner J, Johnston SC, Singhal AB, Becker K, Lansberg MG, Tang W, Kasliwal R, Elkins J. Natalizumab in acute ischemic stroke (ACTION II): A randomized, placebo-controlled trial. Neurology. 2020 Aug 25;95(8):e1091-e1104. doi: 10.1212/WNL.0000000000010038. Epub 2020 Jun 26. PMID 32591475

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 19 sites in Germany, 4 sites in the United Kingdom (UK), 12 sites in Spain, and 18 sites in the United States (US).
Pre-assignment Details: A total of 277 participants with acute ischemic stroke were randomized into the study (94 participants in the placebo group, 91 participants in the natalizumab 300 milligram (mg) group, and 92 participants in the natalizumab 600 mg group).
Groups:
- Placebo: Single dose of matching placebo intravenous (IV) to natalizumab on Day 1 at one of two treatment windows, either within 9 hours or between 9-24 hours from when the participant was last known normal (LKN).
- Natalizumab 300 mg IV: Single 300 mg natalizumab IV on Day 1 at one of two treatment windows, either within 9 hours or between 9-24 hours from when the participant was last known normal (LKN).
- Natalizumab 600 mg IV: Single 600 mg natalizumab IV on Day 1 at one of two treatment windows, either within 9 hours or between 9-24 hours from when the participant was last known normal (LKN).
Period: Overall Study
Arm/Group | Placebo | Natalizumab 300 mg IV | Natalizumab 600 mg IV
Started | 94 | 91 | 92
Safety Population (Participants who had received any study treatment (including complete or incomplete infusion)) | 91 | 90 | 89
Participants Dosed | 91 | 88 | 91
Who Received Total Volume of Study Drug | 90 | 88 | 89
Completed | 81 | 77 | 81
Not Completed | 13 | 14 | 11
Not completed — Death | 5 | 6 | 4
Not completed — Consent withdrawn | 2 | 4 | 1
Not completed — Lost to Follow-up | 3 | 1 | 4
Not completed — Other | 1 | 1 | 2
Not completed — Other | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Natalizumab 300 mg IV | Natalizumab 600 mg IV | Total
Number analyzed (Participants) | 94 | 91 | 92 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (9.54) | 66.1 (10.47) | 65.6 (11.09) | 66.2 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 36 | 37 | 102
  Male | 65 | 55 | 55 | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 7
  Not Hispanic or Latino | 28 | 24 | 24 | 76
  Unknown or Not Reported | 64 | 65 | 65 | 194
Race/Ethnicity, Customized [Number; unit: count of participants]
  Black or African American | 2 | 1 | 1 | 4
  White | 27 | 25 | 25 | 77
  Not Reported Due to Confidentiality Regulations | 64 | 65 | 65 | 194
  Missing | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite Global Measure of Functional Disability Excellent Outcome at Day 90
Description: The composite global measure of functional disability excellent outcome was based on a score of 0 or 1 on the modified Rankin Scale (mRS) and a score of >=95 on the Barthel Index (BI). mRS measures independence, rather than neurological function, with specific tasks pre- and post-stroke. The scale consists of 7 grades, from 0 to 6, with 0 corresponding to no symptoms and 6 corresponding to death. BI consists of 10 items that measure a participant's daily functioning, specifically the activities of daily living and mobility. The items include feeding, moving from wheelchair to bed and returning, grooming, transferring to and from a toilet, bathing, walking on a level surface, going up and down stairs, dressing, and maintaining continence of bowels and bladder. The scores for each of the items are summed to create a total score of 0 to 100. The higher the score, the more "independent" the participant is.
Time Frame: Day 90
Population: Modified Intent-to-Treat (MITT) population: all randomized participants who had received entire infusion of study treatment. Participants who were accidentally enrolled based on conditions that mimicked stroke symptom at presentation were excluded from MITT population. Number analyzed is the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Natalizumab 300 mg IV | Natalizumab 600 mg IV
Number analyzed (Participants) | 90 | 88 | 89
percentage of participants | 54.1 | 41.5 | 39.9
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg IV; Composite Measure: The global odds ratio was based on a linear logistic regression model with baseline National Institute of Health Stroke Scale (NIHSS) category (score 5-15, 16-23), age (<60, 60-69, 70-80), tissue plasminogen activator (tPA) use (yes/no), treatment window (<=9, >9 and <=24hours), thrombectomy (yes/no) and region (Spain, UK/Germany, United States of America [USA]) as covariates and unstructured working correlation structure; Test type: Superiority; p = 0.086, Regression, Logistic; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.38 to 1.07]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 600 mg IV; Composite Measure: The global odds ratio was based on a linear logistic regression model with baseline NIHSS category (score 5-15, 16-23), age (<60, 60-69, 70-80), tPA use (yes/no), treatment window (<=9, >9 and <=24hours), thrombectomy (yes/no) and region (Spain, UK/Germany, USA) as covariates and unstructured working correlation structure; Test type: Superiority; p = 0.031, Regression, Logistic; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.34 to 0.95]

2. Secondary Outcome: Percentage of Participants With Excellent Outcome in mRS Score at Day 90
Description: Excellent mRS is defined as mRS score of 0 or 1. mRS measures independence, rather than neurological function, with specific tasks pre- and poststroke. The scale consists of 7 grades, from 0 to 6, with 0 corresponding to no symptoms and 6 corresponding to death.
Time Frame: Day 90
Population: MITT population: all randomized participants who had received entire infusion of study treatment. Participants who were accidentally enrolled based on conditions that mimicked stroke symptom at presentation were excluded from MITT population. Number analyzed is number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Natalizumab 300 mg IV | Natalizumab 600 mg IV
Number analyzed (Participants) | 86 | 83 | 82
percentage of participants | 41 | 29 | 26
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg IV; The odds ratio was based on a linear logistic regression model with baseline NIHSS category (score 5-15, 16-23), age (<60, 60-69, 70-80), tPA use (yes/no), treatment window (<=9, >9 and <=24hours), thrombectomy (yes/no) and region (Spain, UK/Germany, USA) as covariates and unstructured working correlation structure; Test type: Superiority; p = 0.222, Regression, Logistic; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.35 to 1.28]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 600 mg IV; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.073, Regression, Logistic; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.28 to 1.06]

3. Secondary Outcome: Percentage of Participants With Excellent Outcome in BI Score at Day 90
Description: Excellent BI outcome is defined as a score of >=95. BI consists of 10 items that measure a participant's daily functioning, specifically the activities of daily living and mobility. The items include feeding, moving from wheelchair to bed and returning, grooming, transferring to and from a toilet, bathing, walking on a level surface, going up and down stairs, dressing, and maintaining continence of bowels and bladder. The scores for each of the items are summed to create a total score of 0 to 100. The higher the score, the more "independent" the participant is.
Time Frame: Day 90
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Natalizumab 300 mg IV | Natalizumab 600 mg IV
Number analyzed (Participants) | 86 | 81 | 81
percentage of participants | 67 | 54 | 54
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg IV; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.085, Regression, Logistic; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.29 to 1.08]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 600 mg IV; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.067, Regression, Logistic; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.28 to 1.04]

4. Secondary Outcome: Stroke Impact Scale-16 (SIS-16) Score Using a Repeated Measures Mixed Effects Model at Day 90
Description: The SIS-16 is a 16-item physical dimension instrument that was developed as a brief, stand-alone tool for measuring the physical aspects of stroke recovery. The 16 physical aspects are rated on a 1 to 5 scale as follows: not difficult at all (5), a little difficult (4), somewhat difficult (3), very difficult (2), and could not do at all (1). Total score range is 16 to 80, with higher scores indicating higher levels of health-related quality of life and function.
Time Frame: Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Natalizumab 300 mg IV | Natalizumab 600 mg IV
Number analyzed (Participants) | 84 | 80 | 77
score on a scale | 76.21 (30.783) | 66.96 (35.493) | 68.10 (31.461)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg IV; Treatment and treatment by visit interaction were included in the model as explanatory variables. Baseline NIHSS category (score 5-15, 16-23), tPA use (yes/no), age (<60, 60-69, 70-80), thrombectomy (yes/no), region (Spain, UK/Germany, USA) and treatment window were considered as covariates. An unstructured variance-covariance matrix was used in the model; Test type: Superiority; p = 0.106, Mixed-effects model for repeated measure; Adjusted Mean Difference = -7.7, 95% CI 2-sided [-16.97 to 1.64]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 600 mg IV; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.202, Mixed-effects model for repeated measure; Adjusted Mean Difference = -6.1, 95% CI 2-sided [-15.43 to 3.27]

5. Secondary Outcome: Montreal Cognitive Assessment (MoCA) Score at Day 90
Description: The MoCA is a global cognitive screening test with favorable psychometric properties It screens 8 domains: visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 0 to 30 points; a score of 26 or above is considered normal, <10 (severe cognitive impairment), 10-17 (moderate cognitive impairment) and >=18 (mild cognitive impairment).
Time Frame: Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Natalizumab 300 mg IV | Natalizumab 600 mg IV
Number analyzed (Participants) | 69 | 74 | 69
score on a scale | 21.23 (8.412) | 20.73 (8.141) | 20.90 (8.223)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg IV; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.780, Mixed-effects model for repeated measure; Adjusted Mean Difference = -0.3, 95% CI 2-sided [-2.64 to 1.99]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 600 mg IV; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.622, Mixed-effects model for repeated measure; Adjusted Mean Difference = -0.6, 95% CI 2-sided [-2.89 to 1.73]

6. Secondary Outcome: Change From Baseline in National Institute of Health Stroke Scale (NIHSS) Score at Day 90
Description: The NIHSS is a reliable tool for rapidly evaluating the effects of acute cerebral infarction. A trained observer rates the participant's ability to answer questions and perform activities relating to level of consciousness, language, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, sensory loss, and extinction and inattention (formerly neglect). There are 15 items. Total score ranges from 0 as normal to a maximum possible total severity score of 42 for all items. Higher the score, more the severity. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Natalizumab 300 mg IV | Natalizumab 600 mg IV
Number analyzed (Participants) | 77 | 76 | 71
score on a scale | -6.14 (6.920) | -5.17 (7.937) | -6.28 (6.510)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg IV; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.315, Mixed-effects model for repeated measure; Adjusted Mean Difference = 1.2, 95% CI 2-sided [-1.10 to 3.40]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 600 mg IV; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.542, Mixed-effects model for repeated measure; Adjusted Mean Difference = -0.7, 95% CI 2-sided [-2.96 to 1.56]

7. Secondary Outcome: Number of Participants Experiencing Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Baseline up to Day 90
Population: The safety population was defined as participants who had received any study treatment, including cases of complete or incomplete infusion.
Measure: Number; unit: participants
Arm/Group | Placebo | Natalizumab 300 mg IV | Natalizumab 600 mg IV
Number analyzed (Participants) | 91 | 90 | 89
participants | 84 | 81 | 82

8. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAE)
Description: A SAE is any untoward medical occurrence that at any dose results in death, is a life-threatening event, requires inpatient hospitalization, results in a significant disability/incapacity or congenital anomaly.
Time Frame: Baseline up to Day 90
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Placebo | Natalizumab 300 mg IV | Natalizumab 600 mg IV
Number analyzed (Participants) | 91 | 90 | 89
participants | 19 | 23 | 29

9. Secondary Outcome: Percentage of Participants With Dose Response at Day 90
Description: Percentage of participants with dose response was evaluated in proportion of excellent outcome on mRS and BI.
Time Frame: Day 90
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Natalizumab 300 mg IV | Natalizumab 600 mg IV
Number analyzed (Participants) | 90 | 88 | 89
percentage of participants
  mRS (0, 1): number analyzed (Participants) | 86 | 83 | 82
  mRS (0, 1) | 41 | 29 | 26
  BI (>=95): number analyzed (Participants) | 86 | 81 | 81
  BI (>=95) | 67 | 54 | 54
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg IV vs Natalizumab 600 mg IV; mRS: The Cochran-Armitage trend test of a monotonically increasing dose response in proportion of excellent outcome. Dose levels are log transformed; Test type: Superiority; p = 0.028, Cochran-Armitage trend test
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 300 mg IV vs Natalizumab 600 mg IV; BI: The Cochran-Armitage trend test of a monotonically increasing dose response in proportion of excellent outcome. Dose levels are log transformed; Test type: Superiority; p = 0.049, Cochran-Armitage trend test

ADVERSE EVENTS:
Time Frame: Baseline up to Day 90
Description: The safety population was defined as participants who had received any study treatment, including cases of complete or incomplete infusion.
Arm/Group | Placebo | Natalizumab 300 mg IV | Natalizumab 600 mg IV
All-Cause Mortality (participants affected / at risk) | 5/91 | 6/90 | 4/89
Serious Adverse Events (participants affected / at risk) | 19/91 | 23/90 | 29/89
Other Adverse Events (participants affected / at risk) | 67/91 | 69/90 | 65/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=91) | Natalizumab 300 mg IV (N=90) | Natalizumab 600 mg IV (N=89)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Haemophilus infection (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1
Pneumonia acinetobacter (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0
Septic encephalopathy (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 1
Splenic abscess (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Aortic restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Escherichia test positive (Investigations) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 3 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 2
Cerebral reperfusion injury (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 3
Cytotoxic oedema (Nervous system disorders) | 0 | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 3 | 2
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1
Neurological decompensation (Nervous system disorders) | 1 | 1 | 1
Partial seizures (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Stroke in evolution (Nervous system disorders) | 1 | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 2
Ureteric rupture (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Idiopathic angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic embolus (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=91) | Natalizumab 300 mg IV (N=90) | Natalizumab 600 mg IV (N=89)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 5
Atrial fibrillation (Cardiac disorders) | 8 | 6 | 7
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 1
Constipation (Gastrointestinal disorders) | 18 | 19 | 23
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 6 | 2
Nausea (Gastrointestinal disorders) | 4 | 7 | 6
Vomiting (Gastrointestinal disorders) | 3 | 7 | 1
Fatigue (General disorders) | 5 | 1 | 1
Pain (General disorders) | 3 | 7 | 2
Pyrexia (General disorders) | 11 | 19 | 14
Pneumonia (Infections and infestations) | 3 | 2 | 8
Urinary tract infection (Infections and infestations) | 11 | 14 | 15
Fall (Injury, poisoning and procedural complications) | 5 | 7 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 12 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2
Haemorrhagic transformation stroke (Nervous system disorders) | 4 | 4 | 5
Headache (Nervous system disorders) | 15 | 16 | 20
Agitation (Psychiatric disorders) | 8 | 5 | 0
Anxiety (Psychiatric disorders) | 4 | 2 | 7
Depression (Psychiatric disorders) | 16 | 13 | 10
Insomnia (Psychiatric disorders) | 4 | 11 | 10
Haematuria (Renal and urinary disorders) | 5 | 3 | 3
Urinary retention (Renal and urinary disorders) | 6 | 4 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 1
Hypertension (Vascular disorders) | 6 | 7 | 8
Hypotension (Vascular disorders) | 5 | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT02730455/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT02730455/SAP_001.pdf